CLINICAL TRIAL: NCT06895720
Title: EFFECT OF SELF-MYOFASCİAL RELEASE ON MUSCLE MECHANİCAL PROPERTİES, PERFORMANCE, NEUROMUSCULAR FUNCTİON AND MİNİMİZATİON OF İNJURY RİSK İN YOUNG SOCCER PLAYERS
Brief Title: THE MYOFASCIAL SYSTEM AND MINIMIZING THE RISK OS INJURY IN SPORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Bruno Ferreira Rondon Linhares, Principal Investigator, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-CED/2024
Record Dates: First submitted 2025-03-05; First posted 2025-03-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Sports Injuries; Flexibility; Balance; Jumping Performance; Muscle Tonus; Ranger of Motion; Reactive Strength Index; Muscle Stiffness; Muscle Elasticity
Keywords: Self-myofascial release; Injury prevention; Muscle mechanical properties
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group - Myofascial Self-Release (Experimental): In this group, the following will be evaluated: muscle mechanical properties using the Myoton, flexibility using the sit-and-reach test, dorsiflexion range of motion using the Weight Bearing Lunge Test, motor control using the Y Balance Test, and the reactive strength index using the Myjump App. Myofascial self-release will be performed using a structured roller.
  Interventions: Other: Myofascial Self-Release
- No Intervention: Control Group (No Intervention): Athletes will maintain regular training sessions

INTERVENTIONS:
Other: Myofascial Self-Release — Athletes will be asked to use the myofascial release roller for 2 minutes before training on each of the three muscle groups: anterior and posterior thigh and posterior leg. They will be instructed to roll while applying as much pressure as possible on the roller. For the anterior thigh, the roller will be moved along the entire front part of the thigh; for the posterior thigh, it will be rolled from just below the gluteal region to just above the knee; and for the posterior leg, it will be rolled from just below the knee to just above the heel.
  Other Names: Foam rolling
  Arms: Experimental Group - Myofascial Self-Release

SUMMARY:
The aim of the study is to evaluate the effect of myofascial self-release on muscle mechanical properties, performance, neuromuscular function, and injury risk reduction in young soccer players. The hypothesis is a reduction in the number of injuries in the experimental group, as well as improvements in muscle mechanical properties, performance, and neuromuscular function in young soccer players.The study will be a randomized clinical trial with a convenience sample of approximately 65 male athletes aged between 14 and 18 years, divided into control and experimental groups. Athletes with no history of injury in the three months prior to the study will be included, while those with a history of previous surgery or lower limb fractures in the past five years, or who are undergoing physiotherapy at the time of the study, will be excluded.Muscle mechanical properties (myotonometry), flexibility (sit-and-reach test), ankle dorsiflexion range of motion (Weight Bearing Lunge Test), motor control (Y Balance Test), and the reactive strength index (Myjump App) will be assessed before, immediately after, and at 8 and 16 weeks post-intervention. Myofascial self-release will be performed bilaterally on the quadriceps, hamstrings, and calves for 2 minutes per region, twice a week, using a structured massage roller. All procedures will be demonstrated beforehand during the study.

For the Myoton procedure, the athlete will simply lie in a supine and prone position on the examination table. The athlete will only be asked to remain still in the "face-up" or "face-down" position, feeling only the light contact of the device's probe, which is painless and will be demonstrated beforehand.

In the Y Balance Test, athletes will be asked to balance on one foot atop a grid placed on the floor, with their hands on their hips, and reach as far as possible with the non-supporting leg in three marked directions on the floor, without lifting the heel of the supporting leg.

For the Ankle Range of Motion - Weight Bearing Lunge Test, the athlete will place the tested foot on a measuring tape positioned on the floor and will be instructed to touch their knee to the wall in front of them without lifting the heel of the tested foot. Three attempts will be allowed, and the longest distance from the big toe to the wall will be recorded.

In the Sit-and-Reach Test, the athlete will sit on the floor with bare feet and both legs extended. They will be instructed to keep their hands side by side and try to reach the greatest possible distance on the ruler in front of them by bending forward without bending their legs, holding the position for one second to measure the distance. Three attempts will be allowed, and the greatest distance reached will be recorded.

For ground reaction strength, the athlete will be asked to jump off a 40 cm high box, and as soon as their feet touch the ground, they will be encouraged to jump upward as quickly and as high as possible.

In myofascial self-release, athletes in the experimental group will be asked to use the myofascial release roller for 2 minutes before training on each of the three muscle groups - anterior and posterior thigh and posterior leg. Athletes will be instructed to roll using as much pressure as possible on the roller. For the anterior thigh, they will roll across the entire front part of the thigh; for the posterior thigh, they will roll from just below the gluteal region to just above the knee; and for the posterior leg, they will roll from just below the knee to just above the heel.

ELIGIBILITY:
Inclusion Criteria:

* Athletes at the youth and junior levels
* Registered with the respective football association
* Athletes with no history of injury in the past 3 months

Exclusion Criteria:

* Athletes who failed pre-season medical examinations
* Athletes with a history of previous surgery or lower limb fractures in the last 5 years
* Athletes undergoing physiotherapy rehabilitation at the time of the study
* Athletes participating in another injury prevention program or specific training

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of sports injuries | Until the completion of the studies, an average of 5 months.
  Monitor the incidence of injuries in the control and experimental groups

SECONDARY OUTCOMES:
Evaluate Muscle Mechanical Properties | For a period of 8 and 16 weeks
  Muscle elasticity will be assessed using myotonometry.
Evaluate Muscle Mechanical Properties | For a period of 8 and 16 weeks
  Tone will be assessed using myotonometry.
Evaluate Muscle Mechanical Properties | For a period of 8 and 16 weeks
  Stiffness will be assessed using myotonometry.
Evaluate Neuromuscular Control | For a period of 8 and 16 weeks
  Neuromuscular control will be assessed using the Y Balance Test.
Evaluate Ankle Dorsiflexion Range of Motion | For a period of 8 and 16 weeks
  Ankle dorsiflexion range of motion will be assessed using the Weight-Bearing Test.
Evaluate Flexibility | For a period of 8 and 16 weeks
  Flexibility will be assessed using the Sit and Reach Test.
Evaluate the Reactive Strength Index | For a period of 8 and 16 weeks
  The Reactive Strength Index will be assessed using the MyJump application.
Evaluate the Jump Height | For a period of 8 and 16 weeks
  The Jump Height will be assessed using the MyJump application.
Evaluate the air time after the jump | For a period of 8 and 16 weeks
  The air time after jump will be assessed using the MyJump application.

CONTACTS AND LOCATIONS:
Locations (1):
- Azevedo Coutinho Street No. 5, Fão, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No